CLINICAL TRIAL: NCT00229047
Title: Ischemia and Reperfusion Injury in the Human: An Observational Study
Status: Completed | Type: Observational
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Responsible Party: Dr. T. Forbes, Lawson Health Research Institute
Other Study IDs: R-05-133; 11268E
Record Dates: First submitted 2005-09-27; First posted 2005-09-29 (Estimated); Last update posted 2017-08-25 (Actual); Status verified 2017-08

CONDITIONS: Ischemia
Keywords: Ischemic Preconditioning; Microvascular Perfusion; Inflammation; Ischemia and Reperfusion; Chronic Limb Ischemia
MeSH Terms: conditions — Ischemia; Inflammation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Vein Stripping: Patients undergoing elective varicose vein stripping in our vascular OR. Observe circulation in the exposed soleus/gastrocnemius muscle.

SUMMARY:
We, the researchers at Lawson Health Research Institute, propose to investigate the impact of surgical ischemia and reperfusion on skeletal muscle microcirculation using a hand-held microscope.

DETAILED DESCRIPTION:
We propose to investigate the impact of surgical ischemia and reperfusion on skeletal muscle microcirculation using a hand-held microscope.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing femoral distal bypass procedures for chronic limb ischemia

Exclusion Criteria:

* Any severe comorbid conditions (i.e., chronic obstructive pulmonary disease [COPD])

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing routine and elective varicose vein stripping.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2005-04 (Actual); Primary Completion 2010-12 (Actual); Study Completion 2011-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Amit Badhwar, PhD, Study Director — Scientist; Tom Forbes, MD, Principal Investigator — Vascular Surgeon
Locations (1):
- Lawson Health Research Institute, London, Ontario, Canada